CLINICAL TRIAL: NCT07173790
Title: Indolent Lymphoma: Is "Watch and Wait" Really "Worry and Wait"? A Patient-Reported Outcomes Study
Brief Title: Watch and Wait or Worry and Wait in Indolent Lymphoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea University Anam Hospital (Other); Samsung Medical Center (Other); Catholic Medical Center of Korea (Unknown)
Responsible Party: Principal Investigator, JaMin Byun, Professor of Hematology/Oncology, Seoul National University Hospital
Other Study IDs: H-2508-149-1670
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lymphocytic Leukemia (CLL) / Small Lymphocytic Lymphoma (SLL); Marginal Zone Lymphoma(MZL); Follicular Lymphoma, Grade 1; Follicular Lymphoma, Grade 2; Waldenström Macroglobulinemia (WM); Lymphoplasmacytic Lymphoma
Keywords: Indolent lymphoma; PRO; Watch and Wait; Patient-Reported Outcomes; Quality of Life (QoL); Psychosocial Distress
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational cohort: Patients with indolent lymphoma (CLL/SLL, MZL, FL, WM/LPL) who are recently diagnosed and managed with a watch-and-wait strategy. Participants will complete patient-reported outcome surveys assessing quality of life and psychological distress.
  Interventions: Other: Patient-Reported Outcomes Survey

INTERVENTIONS:
Other: Patient-Reported Outcomes Survey — Participants will complete validated questionnaires including EORTC QLQ-C30, EQ-5D-5L, and disease-specific modules (QLQ-CLL17, QLQ-NHL). Responses will be used to assess quality of life and psychological distress during watchful waiting.

SUMMARY:
Indolent lymphomas, including chronic lymphocytic leukemia/small lymphocytic lymphoma, marginal zone lymphoma, low-grade follicular lymphoma, and Waldenström macroglobulinemia, are slow-growing cancers often managed initially with a watchful waiting strategy. This approach avoids unnecessary side effects of early therapy but may negatively impact patients' quality of life (QoL) due to anxiety, uncertainty, and self-monitoring of symptoms. Previous research has suggested increased distress and greater QoL decline in patients under observation compared to those receiving treatment, despite similar or lower disease burden. Moreover, poor QoL has been shown to independently predict overall survival in non-Hodgkin lymphoma patients. However, there are limited data from Asian populations, where cultural factors, health insurance systems, and treatment access differ significantly. This study will evaluate the impact of watchful waiting on patient-reported QoL among Korean patients with indolent lymphoma, providing evidence specific to this population and healthcare setting.

DETAILED DESCRIPTION:
This is an observational, patient-reported outcomes study of indolent lymphoma patients managed with a watch-and-wait strategy. Eligible participants include adults (≥19 years) diagnosed at Seoul National University Hospital with chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone lymphoma (MZL), follicular lymphoma (FL), or Waldenström macroglobulinemia/lymphoplasmacytic lymphoma (WM/LPL), according to WHO criteria. Patients must be recently diagnosed, currently under observation, and able to understand and complete the survey independently. Patients receiving active systemic therapy or with cognitive impairment precluding self-report are excluded.

The target enrollment is up to 150 participants, estimated based on the number of eligible outpatients seen over a 3-month period. Recruitment will occur during outpatient visits, where physicians will introduce the study. After providing written informed consent, patients will complete validated questionnaires (EORTC QLQ-C30, EQ-5D-5L, and disease-specific modules such as QLQ-CLL17 or QLQ-NHL) to assess quality of life, distress, and emotional well-being. Clinical and demographic data (e.g., age, sex, diagnosis, stage, ECOG, marital status, outpatient interval) will also be collected from medical records. Surveys are expected to take at least 20 minutes and will be completed by patients during outpatient waiting periods.

The study involves no therapeutic intervention and poses no risks beyond minimal psychological burden comparable to daily life or routine clinical assessments. Data will be analyzed descriptively and statistically to evaluate the impact of observation on quality of life and psychosocial outcomes. Unlike prior studies, this investigation will focus on Korean patients, reflecting Asian cultural context, local health insurance structure, and treatment accessibility, thereby providing novel and clinically meaningful insights.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥19 years old.
* Diagnosed with indolent lymphoma (CLL/SLL, MZL, FL, or WM/LPL) at Seoul National University Hospital according to WHO criteria.
* Currently managed with watch-and-wait (no active systemic therapy).
* Able to understand and independently complete the study questionnaires.
* Provide voluntary informed consent.

Exclusion Criteria:

* Receiving active systemic anti-lymphoma therapy at the time of enrollment.
* Cognitive impairment or other condition preventing independent completion of the questionnaire.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with indolent lymphoma (CLL/SLL, MZL, FL, or WM/LPL) at Seoul National University Hospital who are managed with a watch-and-wait strategy and able to provide informed consent and complete patient-reported outcome surveys.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | At enrollment during a routine outpatient visit for patients managed with watch-and-wait; single assessment completed once on the day of enrollment (expected 20-30 minutes).
  Patient-reported quality of life will be measured using the validated European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30), which includes global health status/QoL, functional scales, and symptom items. Scores will be transformed to a 0-100 scale according to the official EORTC scoring manual; higher functional and global health scores indicate better quality of life, whereas higher symptom scores indicate worse symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ja Min Byun, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Korea UniversityKorea University Guro Hospital, Seoul, Guro-gu
  - Seoul National University Hospital, Seoul, Jongno-gu
  - The Catholic University of Korea, Seoul, Seocho-gu

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared in order to protect patient confidentiality, as the dataset contains sensitive clinical and patient-reported information. Only aggregate results will be disseminated through publications and presentations.

REFERENCES:
- [Result] Akkad N, Flowers CR. Patient-Reported Outcome Measures (PROMS) in Lymphoma. Curr Oncol. 2025 May 1;32(5):265. doi: 10.3390/curroncol32050265. PMID 40422524
- [Result] Tsang M, Maurer MJ, Habermann TM, Cerhan JR, Nastoupil LJ, McCaughan G, et al. Longitudinal assessment of quality of life (QoL) among patients with follicular lymphoma (FL) according to frontline management strategy and FLIPI risk: Analysis from the LEO Cohort. Presented at: 65th American Society of Hematology (ASH) Annual Meeting; 2023 Dec 9-12; San Diego, CA. Abstract 188382
- [Result] McCaughan D, Roman E, Sheridan R, Hewison A, Smith AG, Patmore R, Howell DA. Patient perspectives of 'Watch and Wait' for chronic haematological cancers: Findings from a qualitative study. Eur J Oncol Nurs. 2023 Aug;65:102349. doi: 10.1016/j.ejon.2023.102349. Epub 2023 May 13. PMID 37331194